CLINICAL TRIAL: NCT05836116
Title: Evaluation of Lateral and Medial Part Activations of Latissimus Dorsi Muscle During Isometric Exercises in Individuals With Scoliosis
Brief Title: Evaluation of Latissimus Dorsi Muscle During Isometric Exercises in Scoliosis
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Muhammet Ayhan ORAL, Assistant Professor, Kırıkkale University
Other Study IDs: LD activation in Scoliosis
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Scoliosis
Keywords: Scoliosis; Latissimus Dorsi Muscle; EMG; Izometric exercises
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Scoliosis: Humans with scoliosis, between age 18-35
  Interventions: Other: Evaluation of Muscle Activation
- Healthy Group (Control group): Healthy human subjects between age 18-35
  Interventions: Other: Evaluation of Muscle Activation

INTERVENTIONS:
Other: Evaluation of Muscle Activation — Evaluation of Muscle Activation The sEMG device, which is a surface EMG system (Myomonitor, Delsys Inc, Boston, MA), was used to measure the lateral and medial muscle activation levels of the latissimus dorsi.
  Electrode placement was determined according to SENIAM (Surface Electromyography for Non-Invasive Evaluation of Muscles) criteria.
  Evaluation of the Gibbosity Trunk rotation (gibbosity) assessments were performed using Adam's test and using a scoliometer . The bending test (Adam's test) is performed in both standing and forward bending positions. The standing version was used in our study.Each measurement equal to 0° on the scoliometer was defined as symmetry at the measured level of the trunk. All other scoliometer values were defined as asymmetry.
  Evaluation of the Cobb Angle Cobb angles of the curves of the individuals participating in the study were measured with the MicroDicom application.
  Other Names: Evaluation of Cobb Angle; Evaluation of Gibbosity

SUMMARY:
Scoliosis is a complex three-dimensional deformity of the spine, of uncertain etiology, but multifactorial and mainly involves characteristic changes in the sagittal plane also, changes in the coronal plane, and varying degrees of vertebral rotation in the axial plane. In recent studies, pre-scoliotic changes are also examined. Some risk factors for the development of scoliosis include gender, age, ethnicity, and family history. Since apical rotation, gibbosity, and costa vertebral angle are considered to be associated with rotation in the literature, these parameters have been defined as risk factors for the progression of the curve.

Cobb angle, Risser sign, and chronological age are taken as the basis to determine the progression of scoliosis.The onset, progression, and treatment of scoliosis include biomechanical changes and parameters. Structural changes, biomechanical changes, and asymmetries develop between the concave and convex sides. Some studies show that paravertebral muscle asymmetry is caused by the curvature of the spine. Trapeze, LD (latissimus dorsi), and erector spine muscles are examples of paravertebral muscles affected.

The LD is a large, smooth muscle lining the lower posterior rib cage and is one of the paravertebral muscles most commonly affected in scoliosis. LD has shoulder, lumbar spine, and sacroiliac joint connections. Scapula, rib cage, and lumbar region deformities seen in scoliosis can be explained by LD. This may make LD a significant cause of scoliosis. In addition, dynamic and static muscle activation rates of LD should be considered in the diagnosis of scoliosis.In the treatment of scoliosis, treatment methods such as physiotherapeutic scoliosis-specific exercise (PSSE), corset, surgery, EMG biofeedback, and neuromuscular training are used.This asymmetry observed in the paraspinal muscles of individuals with scoliosis made us think that we should analyze the LD muscular activations in more detail. The aim of our study is to examine the muscle activation values of the lateral and medial parts of the LD during isometric exercises.

DETAILED DESCRIPTION:
Scoliosis is a complex three-dimensional deformity of the spine, of uncertain etiology, but multifactorial and mainly involves characteristic changes in the sagittal plane also, changes in the coronal plane, and varying degrees of vertebral rotation in the axial plane. The prevalence of scoliosis in the general population worldwide is 0.93% to 12%. In the last few decades, different factors affecting the prevalence of scoliosis have been identified, such as gender, age, skeletal maturity, body mass index, family history, and ethnicity. Discussions about the causes of scoliosis are still ongoing, whether it is only genetic or due to factors such as exercise and environment. In recent studies, pre-scoliotic changes are also examined. Some risk factors for the development of scoliosis include gender, age, ethnicity, and family history. Since apical rotation, gibbosity, and costa vertebral angle are considered to be associated with rotation in the literature, these parameters have been defined as risk factors for the progression of the curve.

Cobb angle, Risser sign, and chronological age are taken as the basis to determine the progression of scoliosis. The main diagnostic criterion for scoliosis with varying degrees of vertebral axial rotation is spinal curvature greater than or equal to 10° in the coronal plane on a flat anteroposterior X-ray image. The Adam's Test is universally accepted as the primary means of diagnosing scoliosis. The Adam's test shows the rotational component of scoliosis. The onset, progression, and treatment of scoliosis include biomechanical changes and parameters. Structural changes, biomechanical changes, and asymmetries develop between the concave and convex sides. Some studies show that paravertebral muscle asymmetry is caused by the curvature of the spine. Trapeze, LD (latissimus dorsi), and erector spine muscles are examples of paravertebral muscles affected.

The LD is a large, smooth muscle lining the lower posterior rib cage and is one of the paravertebral muscles most commonly affected in scoliosis. LD has shoulder, lumbar spine, and sacroiliac joint connections. Scapula, rib cage, and lumbar region deformities seen in scoliosis can be explained by LD. This may make LD a significant cause of scoliosis. In addition, dynamic and static muscle activation rates of LD should be considered in the diagnosis of scoliosis.

Although guidelines have been established for treatments in the direction of spinal curvature, the choice of treatment type is often subjective and based on clinicians' experience. In the treatment of scoliosis, treatment methods such as physiotherapeutic scoliosis-specific exercise (PSSE), corset, surgery, EMG biofeedback, and neuromuscular training are used. Asymmetry observed in the paraspinal muscles of individuals with scoliosis made us think that we should analyze the LD muscular activations in more detail. The aim of our study is to examine the muscle activation values of the lateral and medial parts of the LD during isometric exercises.

ELIGIBILITY:
Inclusion Criteria:

Scoliosis group

* aged 18-35,
* Risser stage >4,
* Cobb angle of 10-35°,
* range of 18 <BMI <25,
* volunteered to participate

Healthy group

* aged 18-35,
* range of 18 <BMI <25,
* volunteered to participate

Exclusion Criteria:

* with a history of neuromuscular, cardiovascular, pulmonary, vestibular, or rheumatological diseases,
* had previously received any surgical or conservative treatment of the spine,
* exercised regularly

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study, which was designed to evaluate the lateral and medial part muscular activations of the LD muscle during isometric exercises in 20 healthy individuals (8 females, 12 males) and 20 individuals with scoliosis (14 females and 6 males) participated total of 40 individuals.
  In the scoliotic group, scoliosis was diagnosed by radiographic imaging by a specialist, referred to receive exercise therapy participated in the study was included.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Muscle activation | 30 minutes
  Latissimus dorsi muscle activation during izometric exercises
  The measurement unit is mV (millivolt)

SECONDARY OUTCOMES:
Cobb angle | 10 minutes
  Cobb angle of affected part of the columba vertebralis
  The measurement unit is degree.
Gibbosity angle | 5 minutes
  Gibosity angle of affected part of the columba vertebralis
  The measurement unit is degree.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMET AYHAN ORAL, PhD, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kouwenhoven JW, Castelein RM. The pathogenesis of adolescent idiopathic scoliosis: review of the literature. Spine (Phila Pa 1976). 2008 Dec 15;33(26):2898-908. doi: 10.1097/BRS.0b013e3181891751. PMID 19092622
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Slattery C, Verma K. Classifications in Brief: The Lenke Classification for Adolescent Idiopathic Scoliosis. Clin Orthop Relat Res. 2018 Nov;476(11):2271-2276. doi: 10.1097/CORR.0000000000000405. No abstract available. PMID 30179943
- [Background] Trobisch P, Suess O, Schwab F. Idiopathic scoliosis. Dtsch Arztebl Int. 2010 Dec;107(49):875-83; quiz 884. doi: 10.3238/arztebl.2010.0875. Epub 2010 Dec 10. PMID 21191550
- [Background] Liang R, Yip J, Fan Y, Cheung JPY, To KM. Electromyographic Analysis of Paraspinal Muscles of Scoliosis Patients Using Machine Learning Approaches. Int J Environ Res Public Health. 2022 Jan 21;19(3):1177. doi: 10.3390/ijerph19031177. PMID 35162203
- [Background] Castelein RM, Pasha S, Cheng JC, Dubousset J. Idiopathic Scoliosis as a Rotatory Decompensation of the Spine. J Bone Miner Res. 2020 Oct;35(10):1850-1857. doi: 10.1002/jbmr.4137. Epub 2020 Sep 9. PMID 32697856
- [Background] Zhang Y, Yang Y, Dang X, Zhao L, Ren J, Zhang L, Sun J. Factors relating to curve progression in female patients with adolescent idiopathic scoliosis treated with a brace. Eur Spine J. 2015 Feb;24(2):244-8. doi: 10.1007/s00586-014-3674-3. Epub 2014 Nov 26. PMID 25424687